CLINICAL TRIAL: NCT00586391
Title: Phase I Study Of CD19 Chimeric Receptor Expressing T Lymphocytes In B-Cell Non Hodgkin's Lymphoma, Acute Lymphocytic Leukemia, and Chronic Lymphocytic Leukemia
Brief Title: CD19 Chimeric Receptor Expressing T Lymphocytes In B-Cell Non Hodgkin's Lymphoma, ALL & CLL
Acronym: CRETI-NH
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Carlos Ramos, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19384-CRETI-NH; NCT00608270 (obsolete NCT alias)
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: B Cell Lymphoma; Chronic Lymphocytic Leukemia; Acute Lymphocytic Leukemia
Keywords: B cell Lymphoma; Cancer; Chronic Lymphocytic Leukemia; CD19 CHIMERIC RECEPTOR EXPRESSING T LYMPHOCYTES; Acute Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CD19CAR-28-zeta T cells (Experimental): Three dose levels of CTLs will be evaluated. Each patient will receive one injection according to their assigned dose over 1-10 minutes IV.
  *At the discretion of the attending physician, if after a 4 to 6-week evaluation period the patient has had apparent clinical benefit (as determined by symptoms, physical exam or radiological studies); repeat infusions separated by 4 to 6 weeks (up to a maximum of 3 extra doses) of modified T cells at the same dose level or below the patient's original dose can be administered.
  Interventions: Genetic: CD19CAR-28-zeta T cells; Drug: Ipilimumab

INTERVENTIONS:
Genetic: CD19CAR-28-zeta T cells — Intravenous injection
  Dose Level 1:
  CD19CAR-28zeta - 2x10^7 cells/m^2
  Dose Level 2:
  CD19CAR-28zeta - 1 x10^8 cells/m^2
  Dose Level 3:
  CD19CAR-28zeta - 2x10^8 cells/m^2
Drug: Ipilimumab — For patients with intermediate or low grade leukemia/lymphoma, patients may receive ipilimumab once during the week 2 visit after the T cell infusion.
  Other Names: Yervoy

SUMMARY:
Patients on this study have a type of lymph gland cancer called non-Hodgkin Lymphoma, Acute Lymphocytic Leukemia, or chronic Lymphocytic Leukemia (these diseases will be referred to as "Lymphoma" or "Leukemia"). Their Lymphoma or Leukemia has come back or has not gone away after treatment (including the best treatment known for these cancers). This research study is a gene transfer study using special immune cells.

The body has different ways of fighting infection and disease. No one way seems perfect for fighting cancers. This research study combines two different ways of fighting disease, antibodies and T cells, hoping that they will work together. Antibodies are types of proteins that protect the body from bacterial and other diseases. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells including tumor cells. Both antibodies and T cells have been used to treat patients with cancers; they have shown promise, but have not been strong enough to cure most patients.

T lymphocytes can kill tumor cells but there normally are not enough of them to kill all the tumor cells. Some researchers have taken T cells from a person's blood, grown more of them in the laboratory and then given them back to the person.

The antibody used in this study is called anti-CD19. It first came from mice that have developed immunity to human lymphoma. This antibody sticks to cancer cells because of a substance on the outside of these cells called CD19. CD19 antibodies have been used to treat people with lymphoma and Leukemia. For this study anti-CD19 has been changed so that instead of floating free in the blood it is now joined to the T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor.

In the laboratory, investigators have also found that T cells work better if they also put a protein that stimulates T cells called CD28. Investigators hope that adding the CD28 might also make the cells last for a longer time in the body.

These CD19 chimeric receptor T cells with C28 T cells are investigational products not approved by the Food and Drug Administration.

The purpose of this study is to find the biggest dose of chimeric T cells that is safe, to see how the T cell with this sort of chimeric receptor lasts, to learn what the side effects are and to see whether this therapy might help people with lymphoma or leukemia.

DETAILED DESCRIPTION:
Patients will give us blood to make CD19 CD28 chimeric receptor-T cells in the laboratory. These cells will be grown and frozen for the patient. To make the T cells investigators take the blood and stimulate it with growth factors to make the T cells grow. To get the CD19 antibody (with CD28) to attach to the surface of the T cell, they insert the antibody gene into the T cell. This is done with a virus called a retrovirus that has been made for this study and will carry the antibody gene into the T cell. This virus also helps us find the T cells in the blood after they inject them using a special laboratory test. Because the patients will receive cells with a new gene in them they will be followed for a total of 15 years to see if there are any long term side effects of gene transfer. If the patient cannot visit the clinic, they may be contacted by the research coordinator or physician.

When the patients enroll on this study, they will be assigned a dose of CD19 CD28 chimeric receptor-T cells.

For those with intermediate or low grade lymphoma/leukemia: The investigators' studies so far have shown that the infused T cells may need to receive an extra boost in order to expand efficiently in the body. Therefore, 2 weeks after T cell infusion, the patient may receive one injection of a drug called ipilimumab, which they believe will help the T cells grow. This drug is approved by the FDA to treat certain cancers, such as melanoma, but the dose of drug used for this study will be lower than those used in those other treatments to avoid side effects.

Patients will be given an injection of cells into the vein through an IV at the assigned dose. The injection will take about 10 minutes. Patients will be followed in the clinic after the injection for up to 3 hours. If after a 4-6 week evaluation period after the infusion, the patient seems to be experiencing a benefit (confirmed by radiological studies, physical exam and/or symptoms), they may be able to receive up to three additional doses of the T cells if they wish. These additional infusions would be at least 4-6 weeks apart and at the same dose level they received the first time or a lower dose. The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital.

To learn more about the way the CD19 CD28 chimeric receptor-T cells are working and how long they last in the body, extra blood will be drawn.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients must meet the following eligibility criteria to be included:

1. Recurrent B cell lymphoma or leukemia (ALL or CLL), or newly diagnosed patients unable to receive or complete standard therapy OR diagnosis of intermediate B cell lymphoma with a treatment plan that will include high dose therapy and autologous stem cell transplantation. If a patient is less than 18, the lymphoma/leukemia is highly aggressive (i.e. lymphoblastic, Burkitt, ALL).
2. Life expectancy of at least 12 weeks
3. Recovered from the toxic effects of all prior chemotherapy before entering this study
4. ANC greater than 500, HgB greater than 8.0
5. Bilirubin less than 3 times the upper limit of normal
6. AST less than 5 times the upper limit of normal
7. Serum creatinine less than 3 times upper limit of normal
8. Pulse oximetry of greater than 90% on room air
9. Karnofsky/Lansky score of greater than 60%
10. Available autologous transduced peripheral blood T-cells with greater than/=15% expression of CD19CAR determined by flow-cytometry
11. Patients or legal guardians must sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side effects. Patients or their guardians will be given a copy of the consent form
12. Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 3 months after the study is concluded. The male partner should use a condom

EXCLUSION CRITERIA:

1. History of hypersensitivity reactions to murine protein-containing products
2. Pregnant or lactating
3. Tumor in a location where enlargement could cause airway obstruction
4. Currently receiving any investigational agents or have not received any tumor vaccines within the previous six weeks

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-02; Primary Completion 2014-07 (Actual); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Adverse Event Data per Patient | 6 weeks
  Evaluate the safety of autologous T-lymphocytes genetically modified to express CAR targeting CD19CAR in patients with NHL, ALL or B-CLL.

SECONDARY OUTCOMES:
Survival and function of CD19CAR T cells | 15 years
  survival will be measured by a real time Q-PCR assay to detect CD19.CAR T cells in peripheral blood from subjects. Plotts will be generated to depict patterns of survival. Function will be assessed by assays.
Number of patients with tumor response | 6 weeks
  To measure the anti-tumor effects of chimeric CD19 receptor transduced autologous T- lymphocytes in patients with Low-grade non-Hodgkin's Lymphoma (NHL) and Leukemia
Correlation of additional doses and cumulative rise in the percentage of circulating gene modified cells | 15 years
  To discover if the clinical and laboratory data collected following the additional doses of cells are consistent with a cumulative rise in the percentage of circulating gene modified cells and if the infusions are associated with sequential reductions in patient disease burden.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Ramos, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Xu Y, Zhang M, Ramos CA, Durett A, Liu E, Dakhova O, Liu H, Creighton CJ, Gee AP, Heslop HE, Rooney CM, Savoldo B, Dotti G. Closely related T-memory stem cells correlate with in vivo expansion of CAR.CD19-T cells and are preserved by IL-7 and IL-15. Blood. 2014 Jun 12;123(24):3750-9. doi: 10.1182/blood-2014-01-552174. Epub 2014 Apr 29. PMID 24782509